CLINICAL TRIAL: NCT03482791
Title: A Phase II Study of Proton Beam Therapy in the Treatment of Esophageal Cancer
Brief Title: Proton Beam Therapy in the Treatment of Esophageal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201803092
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Esophagus Cancer; Esophageal Cancer; Cancer of the Esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Proton Therapy; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1: Resectable (proton beam therapy) (Experimental): * Proton beam therapy: total dose of 50 or 50.4 Gy
  * Standard of care chemotherapy - the clinical trial doesn't dictate anything about the chemotherapy given, it is the treating physician's decision
  * Surgery should ideally be performed no later than 8 to 10 weeks after completing chemoradiation
  * Patient-reported outcome measures (PROs) performed at several time points
  Interventions: Radiation: Proton beam therapy; Other: Patient-Reported Outcome Measures
- Arm 2: Unresectable (proton beam therapy) (Experimental): * Proton beam therapy: total dose of 59.4 or 60 Gy
  * Standard of care chemotherapy - the clinical trial doesn't dictate anything about the chemotherapy given, it is the treating physician's decision
  * Patient-reported outcome measures (PROs) performed at several time points
  Interventions: Radiation: Proton beam therapy; Other: Patient-Reported Outcome Measures

INTERVENTIONS:
Radiation: Proton beam therapy — * The daily prescription dose will be 1.8 or 2 Gy RBE ("Relative Biologic Equivalence") to be delivered to the periphery of the planning target volume (PTV).
  * The Mevion S-250 Proton Radiation Beam Therapy System will be used.
  Other Names: PBT
Other: Patient-Reported Outcome Measures — -Prior to start of therapy, end of chemoradiation (day of end of treatment or up to 1 week after), 8 weeks, 4, 6, 9, and 12-months following end of chemoradiation
  Other Names: PROs

SUMMARY:
The investigators plan to include both operable and inoperable patients with esophagus cancer in this prospective trial. Since both proton and photon treatments are biologically equivalent, the investigators do not expect a difference in tumor control compared to intensity modulated radiation therapy (IMRT). The investigators have a prospective experience of physician-reported toxicity and patient outcome using IMRT for patients with inoperable esophagus cancer that will serve as a comparison group. For the resectable patients receiving trimodality therapy (chemoradiation followed by surgery), the investigators will carefully track toxicity and patient outcomes prospectively. The central hypothesis is that the biologic efficacy for tumor control should be similar between protons and photons, and therefore survival measures should be similar between the two groups, but that the main difference lies in the total severe toxicities experienced by the patients undergoing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented adenocarcinoma or squamous cell carcinoma of the cervical or thoracic esophagus or gastroesophageal junction or cardia of stomach.
* Staged by PET/CT and esophagogastroduodenoscopy (EGD) or endoscopic ultrasound (EUS) OR CT w/contrast and EGD to have stage II or III disease per AJCC 7th edition guidelines
* Prior endoscopic mucosal resection (EMR) with a diagnosis of stage II or III esophageal cancer (AJCC 7th edition) is eligible, irrespective of margin status.
* Induction chemotherapy prior to concurrent chemoradiation is allowed.
* Prior thoracic radiation is allowable if degree of overlap with the esophageal radiotherapy treatment is deemed to be safe by the treating radiation oncologist.
* At least 18 years of age.
* ECOG performance status < 2
* Normal bone marrow and organ function as defined below:

  * WBC > 2,500/mcL
  * Platelets > 75,000/mcl
  * Total bilirubin < 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) < 3.0 x IULN
  * Creatinine < 1.5 x IULN OR Creatinine clearance > 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.
* English speaker.
* Financial coverage for proton therapy.

Exclusion Criteria:

* Planned treatment with radiation therapy alone without concurrent chemotherapy or chemotherapy alone.
* Previous or concomitant cancers within the past 3 years other than curatively treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, curative treatment for transitional cell carcinoma of the bladder, and low risk prostate cancer. Except for prostate cancer (which can be observed if low risk), other cancers listed must have been treated in the past 3 years without evidence of recurrence at the time of registration.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia not controlled by pacer device, myocardial infarction within 3 months of registration, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 7 days of the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2026-08-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Vlacich, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Started | 16 | 6
Completed | 15 | 6
Not Completed | 1 | 0
Not completed — Patient did not start treatment due to physician decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy) | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Continuous [Median (Full Range); unit: years] | 68.5 [52 to 78] | 77.5 [55 to 84] | 70.5 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 6 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the MD Anderson Symptom Inventory (MDASI)-Plus
Description: The MDASI-Plus is a reliable, validated tool for assessing cancer-related symptoms regardless of therapy or specific cancer diagnosis. Patients are asked to fill out a twenty-seven question inventory. 21 questions ask the patient about the severity of their symptoms with answers ranging from 0=not present to 10=as bad as you can imagine. 6 questions ask the patient about how their symptoms interfered with their life with answers ranging from 0=did not interfere to 10=interfered completely. The higher the score the more severe symptom experience the patient experienced.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 13 | 6
score on a scale
  Baseline: number analyzed (Participants) | 8 | 3
  Baseline | 1.994 (1.641) | 1.127 (0.634)
  Post completion of chemoradiation: number analyzed (Participants) | 6 | 4
  Post completion of chemoradiation | 4.135 (1.795) | 3.024 (2.454)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 1.012 (1) | 1.31 (1.112)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 2.429 (2.107) | 1.714 (2.603)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 1 (0.632) | 0.738 (1.044)

2. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the EuroQol (EQ-5D) Questionnaire
Description: The EQ-5D is a standardized 2-part, patient-administered instrument used for direct and indirect assessment of health state utilities. The first part asks respondents to "check the ONE box [next to the appropriate statement] that best describes your health TODAY" for each of 5 health dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The second part of the EQ-5D is a visual analogue scale (VAS) valuing current health state. Both the 5-item index score and the VAS score are transformed into a utility score between 0 "Worst health state" and 1 "Best health state. The higher the score the better health a patient experienced.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 15 | 6
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 0.664 (0.405) | 0.486 (0.496)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 0.56 (0.358) | 0.607 (0.39)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 0.803 (0.295) | 0.818 (0.124)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 0.802 (0.287) | 0.645 (0.488)
  6 months: number analyzed (Participants) | 8 | 2
  6 months | 0.816 (0.202) | 0.942 (0.083)

3. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the Medical Outcomes Study (MOS) Social Support Survey
Description: The 19-item MOS Social Support Survey was designed for use with patients with chronic diseases and measures how often different kinds of support are available, if needed. Response choices range from "none of the time" (1) to "all of the time" (5). A mean social support score for all 19 items is computed to a 0-100 scale with higher scores indicating a greater availability of social support.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 14 | 6
score on a scale
  Baseline: number analyzed (Participants) | 9 | 4
  Baseline | 89 (14.2) | 71.1 (25.8)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 88.2 (15.8) | 83.4 (24.4)
  2 months: number analyzed (Participants) | 7 | 4
  2 months | 90.2 (15.9) | 98.4 (3.3)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 88.5 (25.3) | 84.2 (27.3)
  6 months: number analyzed (Participants) | 8 | 2
  6 months | 88.2 (16.8) | 98.7 (1.9)

4. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the 4-Item Center for Epidemiological Studies Depression Scale (CES-D)
Description: The CES-D questionnaire is a 20-item measure which evaluates depressive symptoms. This trial will make use of the validated 4-item screening version in order to reduce participant burden. Possible range of scores is 0-60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 15 | 6
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 19.763 (13.438) | 16.355 (11.098)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 4
  Post completion of chemoradiation | 16.67 (7.287) | 15.914 (11.118)
  2 months: number analyzed (Participants) | 7 | 4
  2 months | 12.47 (4.758) | 14.15 (8.316)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 12.47 (5.845) | 14.15 (10.184)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 11.21 (5.368) | 11.21 (4.158)

5. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the MD Anderson Symptom Inventory (MDASI)-Plus
Description: as for outcome 1
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 14 | 6
score on a scale
  Baseline: number analyzed (Participants) | 8 | 3
  Baseline | 1.994 (1.641) | 1.127 (0.634)
  Post completion of chemoradiation: number analyzed (Participants) | 6 | 4
  Post completion of chemoradiation | 4.135 (1.795) | 3.024 (2.454)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 1.012 (1) | 1.31 (1.112)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 2.429 (2.107) | 1.714 (2.603)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 1 (0.632) | 0.738 (1.044)
  9 months: number analyzed (Participants) | 7 | 1
  9 months | 0.878 (0.858) | 2.476
  12 months: number analyzed (Participants) | 7 | 2
  12 months | 1.224 (1.319) | 0.524 (0.202)

6. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the EuroQol (EQ-5D) Questionnaire
Description: as for outcome 2
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 15 | 6
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 0.664 (0.405) | 0.486 (0.496)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 0.56 (0.358) | 0.607 (0.39)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 0.803 (0.295) | 0.818 (0.124)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 0.802 (0.287) | 0.645 (0.488)
  6 months: number analyzed (Participants) | 8 | 2
  6 months | 0.816 (0.202) | 0.942 (0.083)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 0.863 (0.161) | 0.734 (0.377)
  12 months: number analyzed (Participants) | 9 | 2
  12 months | 0.84 (0.181) | 1 (0)

7. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the Medical Outcomes Study (MOS) Social Support Survey
Description: as for outcome 3
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 14 | 6
score on a scale
  Baseline: number analyzed (Participants) | 9 | 4
  Baseline | 89.0 (14.2) | 71.1 (25.8)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 4
  Post completion of chemoradiation | 88.2 (15.8) | 83.4 (24.4)
  2 months: number analyzed (Participants) | 7 | 4
  2 months | 90.2 (15.9) | 98.4 (3.3)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 88.5 (25.3) | 84.2 (27.3)
  6 months: number analyzed (Participants) | 8 | 2
  6 months | 88.2 (16.8) | 98.7 (1.9)
  9 months: number analyzed (Participants) | 6 | 2
  9 months | 87.5 (18.8) | 99.3 (0.9)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 91.8 (11.3) | 100 (0)

8. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the 4-Item Center for Epidemiological Studies Depression Scale (CES-D)
Description: as for outcome 4
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 15 | 6
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 19.763 (13.438) | 16.355 (11.098)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 16.67 (7.287) | 15.914 (11.118)
  2 months: number analyzed (Participants) | 7 | 4
  2 months | 12.47 (4.758) | 14.15 (8.316)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 12.47 (5.845) | 14.15 (10.184)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 11.21 (5.368) | 11.21 (4.158)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 12.89 (5.052) | 8.27 (0)
  12 months: number analyzed (Participants) | 9 | 2
  12 months | 12.843 (5.323) | 8.27 (0)

9. Primary Outcome: Physician-reported Toxicity of PBT for Esophageal Cancer
Description: Number of participants with grade 3 or higher specific cardiac, metabolism/nutrition, gastrointestinal, respiratory/thoracic/mediastinal, and skin/subcutaneous toxicity using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 related to PBT
Time Frame: Through 6 months following chemoradiation (estimated to be 9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 15 | 6
Participants | 2 | 0

10. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Mental Component Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher scores indicate better quality of life.
  MCS scores from the SF-12 are recoded, weighted, and summed, and standardized by the SF-12 scoring procedure. SF-12 is a licensed product and this procedure is implemented in the QualityMetric PRO CoRE software package. MCS range is 40-65.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 45.0 (15.1) | 44.5 (16.4)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 45.7 (9.6) | 45.7 (13.0)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 50.9 (11.0) | 45.3 (15.9)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 50.4 (10.2) | 44.6 (12.3)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 50.8 (8.2) | 54.7 (1.4)

11. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Physical Component Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher scores indicate better quality of life.
  PCS scores from the SF-12 are recoded, weighted, and summed, and standardized by the SF-12 scoring procedure. SF-12 is a licensed product and this procedure is implemented in the QualityMetric PRO CoRE software package. PCS range is 30-55.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, and 6 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 45.8 (12.6) | 41.9 (18.1)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 33.5 (10.5) | 37.6 (11.4)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 40.4 (12.0) | 39.4 (12.6)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 42.6 (13.3) | 42.9 (14.2)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 42.3 (12.0) | 51.9 (6.1)

12. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Physical Component Score
Description: as for outcome 11
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 45.8 (12.6) | 41.9 (18.1)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 33.5 (10.5) | 37.6 (11.4)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 40.4 (12.0) | 39.4 (12.6)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 42.6 (13.3) | 42.9 (14.2)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 42.3 (12.0) | 51.9 (6.1)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 43.9 (9.8) | 40.4 (17.6)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 42.1 (11.1) | 39.8 (7.2)

13. Secondary Outcome: Progression-free Survival (PFS) of Proton Beam Therapy (PBT) for Patients With Resectable
Description: -PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: 5 years following chemoradiation (estimated to be 5 years and 3 months)
Reporting Status: Not Posted, anticipated posting 2027-08

14. Secondary Outcome: Overall Survival (OS)of PBT for Patients With Resectable Versus Unresectable Esophageal
Time Frame: 5 years following chemoradiation (estimated to be 5 years and 3 months)
Reporting Status: Not Posted, anticipated posting 2027-08

15. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Mental Component Score
Description: as for outcome 10
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 45.0 (15.1) | 44.5 (16.4)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 45.7 (9.6) | 45.7 (13.0)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 50.9 (11.0) | 45.3 (15.9)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 50.4 (10.2) | 44.6 (12.3)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 50.8 (8.2) | 54.7 (1.4)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 48.2 (8.6) | 47.9 (16.0)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 51.6 (7.9) | 61.4 (5.3)

16. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - General Health Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Lower mean scores indicate better quality of life.
  The subscales are calculated by recoding and averaging the raw scores (Likert scales) the questions associated with the subscale. Range of 1-5.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 3 (1.3) | 3.5 (1.9)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 3.1 (0.9) | 2.8 (1.1)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 2.5 (0.8) | 3.2 (1.5)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 3 (0.8) | 3 (1)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 3.1 (1.1) | 2.5 (0.7)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 3.1 (0.9) | 3 (1.4)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 3.1 (1) | 2 (0)

17. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Physical Function Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher mean scores indicate better quality of life.
  The subscales are calculated by recoding and averaging the raw scores (Likert scales) the questions associated with the subscale. Range of 1-3.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 2.6 (0.7) | 2.6 (0.7)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 1.9 (0.6) | 1.7 (0.8)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 2.1 (0.8) | 1.9 (0.8)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 2.2 (0.7) | 2.2 (1)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 2.4 (0.6) | 2.5 (1)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 2.3 (0.6) | 1.8 (1)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 2.4 (0.8) | 1.8 (0.5)

18. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Physical Role Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher mean scores indicate better quality of life.
  The subscales are calculated by recoding and averaging the raw scores (Likert scales) the questions associated with the subscale. Range of 1-2.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 1.5 (0.5) | 1.5 (0.5)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 1.1 (0.4) | 1.3 (0.5)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 1.5 (0.5) | 1.2 (0.5)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 1.5 (0.5) | 1.3 (0.5)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 1.5 (0.5) | 2 (0)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 1.5 (0.5) | 1.5 (0.6)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 1.5 (0.5) | 1.5 (0.6)

19. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Emotional Role Score
Description: as for outcome 18
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 1.6 (0.5) | 1.8 (0.5)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 1.6 (0.5) | 1.5 (0.5)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 1.7 (0.5) | 1.5 (0.5)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 1.5 (0.5) | 1.3 (0.5)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 1.8 (0.4) | 2 (0)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 1.6 (0.5) | 1.5 (0.6)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 1.8 (0.4) | 2 (0)

20. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Bodily Pain Score
Description: as for outcome 16
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 2.1 (1.3) | 2.5 (1.9)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 3.1 (1.2) | 2 (1.2)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 2.6 (1.5) | 1.5 (1)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 2 (1.5) | 1.7 (1.2)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 1.9 (1.1) | 1 (0)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 1.6 (0.5) | 2 (1.4)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 2 (1.1) | 1.5 (0.7)

21. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Mental Health Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Lower mean scores indicate better quality of life.
  The subscales are calculated by recoding and averaging the raw scores (Likert scales) the questions associated with the subscale. Range of 1-6.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 2.8 (1.4) | 2.8 (1.5)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 2.9 (1.1) | 2.7 (1.3)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 2.1 (1.0) | 2.6 (1.6)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 1.9 (0.9) | 2.5 (1.4)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 2.1 (1.4) | 2.2 (1.0)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 2.5 (1.0) | 2.8 (2.2)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 2.1 (1.0) | 1.5 (0.6)

22. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Vitality Health Score
Description: as for outcome 21
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 3.5 (1.5) | 4 (2.3)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 4.4 (1) | 4.4 (1.5)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 3.4 (1.1) | 4.2 (1.5)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 3.6 (1.7) | 3.7 (1.5)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 3.6 (1.6) | 3 (1.4)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 3.1 (1.5) | 3.5 (2.1)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 3.4 (1.5) | 3 (1.4)

23. Primary Outcome: Change in Patient-reported Outcomes of PBT for Esophageal Cancer as Measured by the SF-12 Questionnaire - Social Functioning Score
Description: The SF-12 will be measured at each of 7 interviews, and mental and physical component scores will be calculated in addition to calculating the measure's eight individual subscales (physical functioning, social functioning, role limitations due to physical problems, body pain, general health, role limitations due to emotional problems general health, vitality, and mental health). Higher mean scores indicate better quality of life.
  The subscales are calculated by recoding and averaging the raw scores (Likert scales) the questions associated with the subscale. Range of 1-5.
Time Frame: Baseline, post completion of chemoradiation, 2 months, 4 months, 6 months, 9 months, and 12 months
Population: Participants who did not complete the questionnaires are not included in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
Number analyzed (Participants) | 11 | 5
score on a scale
  Baseline: number analyzed (Participants) | 11 | 4
  Baseline | 3.9 (1.4) | 3 (1.8)
  Post completion of chemoradiation: number analyzed (Participants) | 7 | 5
  Post completion of chemoradiation | 2.9 (1.3) | 3.4 (1.3)
  2 months: number analyzed (Participants) | 8 | 4
  2 months | 3.6 (1.4) | 3.8 (1)
  4 months: number analyzed (Participants) | 7 | 3
  4 months | 4.3 (1.3) | 3.7 (1.5)
  6 months: number analyzed (Participants) | 7 | 2
  6 months | 4 (1.2) | 5 (0)
  9 months: number analyzed (Participants) | 7 | 2
  9 months | 3.9 (1.3) | 4 (1.4)
  12 months: number analyzed (Participants) | 8 | 2
  12 months | 4 (1.1) | 4.5 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from start of treatment through 1 year. All-cause mortality is collected from start of treatment through 5 years.
Arm/Group | Arm 1: Resectable (Proton Beam Therapy) | Arm 2: Unresectable (Proton Beam Therapy)
All-Cause Mortality (participants affected / at risk) | 8/15 | 4/6
Serious Adverse Events (participants affected / at risk) | 12/15 | 4/6
Other Adverse Events (participants affected / at risk) | 5/15 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Resectable (Proton Beam Therapy) (N=15) | Arm 2: Unresectable (Proton Beam Therapy) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Chest pain-cardiac (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericardial tamponade (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
COVID-19 infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
ACE induced cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery pseudoaneurysm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Resectable (Proton Beam Therapy) (N=15) | Arm 2: Unresectable (Proton Beam Therapy) (N=6)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03482791/Prot_SAP_000.pdf